CLINICAL TRIAL: NCT00144196
Title: A 12-week Double-blind, Randomised, Parallel-group, Multi-centre Study Evaluating the Efficacy of Tiotropium Versus Placebo in Patients With Mild COPD, According to Swedish Guidelines (SPIRIMILD)
Brief Title: 12 Week Efficacy of Tiotropium Versus Placebo in Patients With Mild COPD According to Swedish Guidelines (SPIRIMILD)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 205.281
Record Dates: First submitted 2005-09-02; First posted 2005-09-05 (Estimated); Last update posted 2023-12-05 (Actual); Status verified 2023-11

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide

INTERVENTIONS:
Drug: tiotropium (Spiriva)

SUMMARY:
To show that treatment with tiotropium inhalation capsules (18 μg q.d.) via HandiHaler® improves lung function in patients with mild COPD according to Swedish guidelines.

DETAILED DESCRIPTION:
Following an initial screening at the screening visit(Visit 1), patients enter a 2 week run-in period. Patients are allowed to take salbutamol (Ventoline, Diskus, 0.2 mg) prn as rescue medication and have to record their daily use of it on the Patient's Diary. Patients who meet all inclusion and none of the exclusion criteria at the check at Visit 2 will be randomised thereafter into the randomised treatment period of the study during which they will receive either tiotropium(Spiriva) or placebo in blinded fashion.

On Day 0 (Visit 2), the first administration of blinded study medication (tiotropium(Spiriva) or matching placebo) will be performed at the study site, after a pre-dose pulmonary function test (PFT) has been carried out. First administration of blinded study medication will be monitored by the investigator. Post dose PFTs will be performed at 30 min, 1 and 2 hours.

On Days 1 to 83 except Day 14, the blinded study medication will be self-administered by the patients at home. The patients will inhale one capsule (tiotropium)(Spiriva) or matching placebo) using the HandiHaler device once daily in the morning. The morning dose of the blinded study medication should be taken at approximately the same time each morning between 7:00 a.m. and 10:00 a.m.

At visit 3 and 4 PFTs will be performed predose and post dose at 30 minutes, 1 and 2 hours

Study Hypothesis:

The rationale of the study is to show that treatment with tiotropium (Spiriva) 18 ?g inhalation capsule via HandiHaler once daily improves FEV1 when compared with placebo in patients with mild COPD according to Swedish guidelines, i.e., a post-bronchodilator FEV1 < 60% of predicted normal and FEV1 < 70% of FVC.

Comparison(s):

One group will be treated with inhalation powder capsules of tiotropium (Spiriva), 18 micrograms once daily. The other group will be treated with matching placebo. Randomisation is 1:1

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have signed an written informed consent consistent with ICH GCP guidelines and local legislations prior to participation in the trial.
2. Patients with a diagnosis of COPD. COPD is defined as a disease state characterised by the presence of airflow obstruction often due to chronic bronchitis or emphysema; the airflow obstruction is generally progressive, may be accompanied by airway hyperreactivity, and may be partially reversible.
3. Patients 40 years of age or older without any restriction to sex.
4. Patients who currently smoke or who are ex-smokers with a cigarette smoking history of >10 pack-years.
5. Patients who have a relatively stable airway obstruction (at least 4 weeks free of COPD exacerbations) with a post bronchodilator FEV1 ? 60% of predicted normal, a post bronchodilation FEV1 < 70% of FVC, and a MRC symptom score minimum of 2 at Visit 1

Exclusion Criteria:

1. Patients with a history of asthma, allergic rhinitis, atopy, or who have a total (absolute) blood eosinophil count ? 600 per mm3 (= 0.6 * 109/L) of the first determination at Visit 1
2. Patients with known moderate or severe renal insufficiency.
3. Patients with a recent history (i.e., 6 months or less prior to Visit 1) of myocardial infarction.
4. Patients with any unstable or life threatening cardiac arrhythmia, including patients with a newly diagnosed, clinically relevant arrhythmia on the electrocardiogram (ECG) performed at Visit 1 as well as patients with cardiac arrhythmia requiring an intervention (i.e., hospitalisation, cardioversion, pacemaker placement, and automatic implantable cardiac defibrillator (AICD) placement) or a change in drug therapy during the last year prior to Visit 1.
5. Patients who regularly use oxygen therapy.
6. Patients with known active tuberculosis.
7. Patients with a history of cancer within the last 5 years. Patients with treated basal cell carcinoma are allowed.
8. Patients with a history of life threatening pulmonary obstruction or a history of cystic fibrosis or clinically evident bronchiectasis.
9. Patients who have undergone thoracotomy with pulmonary resection.
10. Patients who are currently in a pulmonary rehabilitation program or who have completed a pulmonary rehabilitation program in the 6 weeks prior to the screening visit (Visit 1).
11. Patients with known hypersensitivity to anticholinergic drugs, lactose or any other components of the inhalation capsule delivery system.
12. Patients with known symptomatic hyperplasia or bladder neck obstruction. Patients being treated for prostatic hyperplasia and report minimal symptoms may be included and should continue their medications.
13. Patients with known narrow-angle glaucoma.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224
Dates: Start 2004-03-11 (Actual); Primary Completion 2005-07-25 (Actual); Study Completion 2005-07-25 (Actual)

PRIMARY OUTCOMES:
The primary efficacy endpoint is defined as area under the curve of change in FEV1 from baseline for the time period from pre-dose to 2 hours post dose (AUC0 2hFEV1) after 12 weeks of randomised treatment. | week 12

SECONDARY OUTCOMES:
Change in trough FEV1 from baseline after 12 weeks of randomized treatment | week 12
Change in trough FEV1 % of predicted after 12 weeks of randomized treatment | week 12
AUC0-2h (FEV1 % of predicted) after 12 weeks of randomized treatment | week 12
Change in trough forced vital capacity (FVC) from baseline after 12 weeks of randomized treatment | week 12
AUC0-2hFVC after 12 weeks of randomized treatment | week 12
Weekly average number of doses of rescue therapy used in the daytime, at nighttime, and total daily | week 12
Change in Baseline Dyspnea Index (BDI) scores (R96-2117) | week 12
Change in health related quality of life (HRQoL) scores according to EQ 5D (R96-2382) | week 12
Change of symptom score according to Medical Research Council (MRC) scale | week 12
Change in smoking status | week 12
Change in working status | week 12
Incidences of adverse events | week 2, 12
Pulse rate measured just before spirometry | week 2, 12
systolic blood pressure, measured just before spirometry | week 2, 12
diastolic blood pressure, measured just before spirometry | week 2, 12

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — B.I. Sweden AB
Locations (25):
- Sweden (25):
  - Boehringer Ingelheim Investigational Site, ?tvidaberg
  - Boehringer Ingelheim Investigational Site, Alvesta
  - Boehringer Ingelheim Investigational Site, Boden
  - Boehringer Ingelheim Investigational Site, Dalum
  - Boehringer Ingelheim Investigational Site, Gislaved
  - Boehringer Ingelheim Investigational Site, Gothenburg
  - Boehringer Ingelheim Investigational Site, Hässelby
  - Boehringer Ingelheim Investigational Site, Helsingborg
  - Boehringer Ingelheim Investigational Site, Höllviken
  - Jakobsbergs sjukhus, Birgittavagen 4, Jarfalla
  - Boehringer Ingelheim Investigational Site, Kalmar
  - Boehringer Ingelheim Investigational Site, Karlstad
  - Boehringer Ingelheim Investigational Site, Kristianstad
  - Boehringer Ingelheim Investigational Site, Linköping
  - Boehringer Ingelheim Investigational Site, Lule?
  - KvartersAkuten, Timmermansgatan 26, Lule?
  - Boehringer Ingelheim Investigational Site, Lund
  - Boehringer Ingelheim Investigational Site, Motala
  - Boehringer Ingelheim Investigational Site, Skärholmen
  - Boehringer Ingelheim Investigational Site, Stockholm
  - Halsocentralen, Hans?kervagen 1A, Stugun
  - Alno V?rdcentral, Raholmsvagen 24, Sundsvall
  - Boehringer Ingelheim Investigational Site, Sunne
  - Boehringer Ingelheim Investigational Site, Ulricehamn
  - Boehringer Ingelheim Investigational Site, Uppsala